CLINICAL TRIAL: NCT01040546
Title: The Association of Obesity With Food Intake and Metabolic Syndrome in Adult Aged 40 and Over and the Effect of a Diet- and Exercise- Related Weight Control Intervention Program on Obesity
Brief Title: The Effect of a Diet- and Exercise- Related Weight Control Intervention Program on Obesity in Adult Aged 40 and Over
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Cheng-Chieh Lin, Ph.D., China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DOH97-TD-F-113-96002
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Obesity; Metabolic syndrome; Weight control educational intervention; Food intake
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized education (Experimental): Individualized consultation of health problem, dietary intake and exercise
  Interventions: Behavioral: Individualized education
- Grouped education (Experimental): Grouped consultation of health problem, dietary intake and exercise
  Interventions: Behavioral: Grouped education

INTERVENTIONS:
Behavioral: Individualized education — We conducted a randomized controlled trial to evaluate the effects of three types of weight control educational intervention programs. Obese subjects were randomly allocated into "individualized health education group", "group weight control education" and "mail-delivered health education group".Obese subjects who were randomly allocated into "individualized health education group" received consulting services provided by a doctor, nutritionist and fitness expert. The interventions were 12 sessions over 6 months.
  Arms: Individualized education
Behavioral: Grouped education — We conducted a randomized controlled trial to evaluate the effects of three types of weight control educational intervention programs. Obese subjects were randomly allocated into "individualized health education group", "group weight control education" and "mail-delivered health education group".Obese subjects who were randomly allocated into "grouped health education group" attended 12 sessions of group intervention over 6 months.
  Arms: Grouped education

SUMMARY:
The purpose of this study is to assess study subjects' adherence to different weight control intervention programs and the effect of intervention programs on physical and biochemical examinations, physical fitness, food intake and exercise behaviors and the prevalence of metabolic syndrome and its components' abnormalities.

DETAILED DESCRIPTION:
Obesity and metabolic syndrome increase the risk of developing cardiovascular disease. Besides, they prevail around the world and certainly become the most important health problems globally. Dietary intake and exercise are regarded as the first line approach to reduce the occurrence of obesity and metabolic syndrome. The purpose of this study is to assess study subjects' adherence to different weight control intervention programs and the effect of intervention programs on physical and biochemical examinations, physical fitness, food intake and exercise behaviors and the prevalence of metabolic syndrome and its components' abnormalities.

This is a two-year project. In the first year, we estimated the prevalence of obesity and metabolic syndrome and explored their relationship with dietary intake and exercise status using the cross-sectional framework in subjects aged 40 years and over from Taichung Community Health Study. Then, we conducted a randomized controlled trial to evaluate the effects of three types of weight control educational intervention programs. Obese subjects were randomly allocated into "individualized health education group", "fellowship health education group" and "mail-delivered health education group". The sample size for these three groups was 79, 81, 80, respectively. All subjects received one of three 6-month interventions and were followed up for 1 year and were assessed at 6-month interval.

This study adopted the criteria of WHO for Asia area and the Department of Health (DOH), Executive Yuan, Taiwan to define the obesity. The prevalence of obesity for WHO definition modified for Asians and DOH among Taichung residents aged forty years old and over is 37.34% and 18.79%, respectively. For the effectiveness of weight control educational programs, after 6-month intervention, reductions in weight, BMI, waist, hip, arm, and bad diet habit were observed in all groups. And after 6-month intervention, reductions in BMI is significantly greater in the individualized and fellowship weight control groups than in the "health education group". After 6-month educational intervention, metabolic syndrome in the individualized and fellowship health education groups decreased from 78.48% and 72.84% to 60.76% and 61.73%, respectively, which corresponded to reductions of 17.72% and 11.11% of baseline metabolic syndrome.

Our study's findings indicate that individualized and fellowship health education groups modify food intake and exercise behaviors, and further reduce body composition, level of biomarkers and prevalence of metabolic syndrome and its components abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Those with overweight or central obesity (body mass index >= 24 kg/m2) and/or waist circumference >= 90 cm in men or >= 80 cm in women.

Exclusion Criteria:

* Those with impaired hearing,
* Those who are handicap,
* Those living outland,
* Those who are older than 75 years old, and
* Those participates that cannot keep to regular follow-up in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Weight, BMI, total body fat and waist circumference | 3,6 and 12 months since intervention

SECONDARY OUTCOMES:
Metabolic syndrome and its components | 3,6 and 12 months since intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chieh Lin, Ph.D., Study Chair — China Medical University Hospital
Locations (1):
- Department of Famility Medicine,China Medical University Hospital, Taichung, Taiwan